CLINICAL TRIAL: NCT04866849
Title: The Effect of Bruxism on Temporomandibular Disorders
Status: Completed | Type: Observational
Sponsor: Yerkoy State Hospital (Other)
Responsible Party: Principal Investigator, Başak Çiğdem Karaçay, Spesialist, Yerkoy State Hospital
Other Study IDs: 2017-KAEK-189_2021.03.10_19
Record Dates: First submitted 2021-04-26; First posted 2021-04-30 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Bruxism; Temporomandibular Disorder
Keywords: bruxism; Temporomandibular Disorder
MeSH Terms: conditions — Bruxism; Temporomandibular Joint Disorders | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- STUDY GROUP: patient diagnosed with bruxism The presence of bruxism was based on self-reported bruxism and examination. Self reported bruxism was recorded as "yes" or "no" . Participants were examined for the existence of four clinical signs of bruxism: (I) abnormal tooth wear, (II) impressions of teeth in the buccal area, (III) impressions of teeth on the tongue, and (IV) hypertrophy of the masseter muscle. In this study, clinical signs of bruxism were considered present if one of the four items was answered "yes."
  Interventions: Other: examination
- CONTROL GROUP: healthy volunteers
  Interventions: Other: examination

INTERVENTIONS:
Other: examination — The presence of bruxism was based on self-reported bruxism and examination. Self reported bruxism was recorded as "yes" or "no" . Participants were examined for the existence of four clinical signs of bruxism: (I) abnormal tooth wear, (II) impressions of teeth in the buccal area, (III) impressions of teeth on the tongue, and (IV) hypertrophy of the masseter muscle. In this study, clinical signs of bruxism were considered present if one of the four items was answered "yes."

SUMMARY:
This case-control study consists of 120 participants aged between 18 and 65 years. Case group included 60 patients with bruxism who presented to physical medicine and rehabilitation outpatient clinic between May 2021 and August 2021. Control group included 60 healthy participant. Patients who had temporomandibular region surgery, congenital teporomandibular joint pathologies, and previous temporomandibular region trauma were also excluded. Assessments including age, gender, body mass index (BMI), education level, and symptom duration were recorded. Patients was evaluated according to the Diagnostic Criteria for Temporomandibular Disorders: Assessment Instruments. Patients was evaluated by Diagnostic Criteria for Temporomandibular Disorders: TMD Pain Screener, Symptom questionnaire, Clinical Examination Form from Assessment Instruments Axis I. Pain Drawing, Graded Chronic Pain (version 2), Jaw Functional Limitation Scale-8 (JFLS-8), Patient Health Questionnaire (PHQ-4) , Oral Behaviors Checklist were applied within the scope of Axis II.

DETAILED DESCRIPTION:
The aim of this study was to effect of bruxism on temporomandibular disorders (TMD) diagnosed by means of the research diagnostic criteria for temporomandibular disorders (RDC/TMD).

This case-control study consists of 120 participants aged between 18 and 65 years. Case group will be included 60 patients with bruxism who presented to physical medicine and rehabilitation outpatient clinic between May 2021 and August 2021. Control group will be included 60 healthy participant. Patients who had temporomandibular region surgery, congenital teporomandibular joint pathologies, and previous temporomandibular region trauma were also excluded.

Assessments including age, gender, body mass index (BMI), education level, and symptom duration will be recorded. Patients will evaluated according to the Diagnostic Criteria for Temporomandibular Disorders: Assessment Instruments. Patients was evaluated by Diagnostic Criteria for Temporomandibular Disorders: TMD Pain Screener, Symptom questionnaire, Clinical Examination Form from Assessment Instruments Axis I. Pain Drawing, Graded Chronic Pain (version 2), Jaw Functional Limitation Scale-8 (JFLS-8), Patient Health Questionnaire (PHQ-4) , Oral Behaviors Checklist will applied within the scope of Axis II.

ELIGIBILITY:
Inclusion Criteria:

* Sixty patients diagnosed with bruxism according to self-reported bruxism and examination.
* Sixty healthy volunteers

Exclusion Criteria:

* Patients with temporomandibular region surgery
* Congenital teporomandibular joint pathologies
* Previous temporomandibular region trauma were excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This case-control study consists of 120 participants aged between 18 and 65 years. Case group included 60 patients with bruxism who presented to physical medicine and rehabilitation outpatient clinic between May 2021 and August 2021. Control group included 60 healthy participant.
Sampling Method: Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-08-25 (Actual)

PRIMARY OUTCOMES:
DCTMD: AI Axis I Pain Screener | 0 day
  MD Pain Screener which is a simple, reliable, and valid self-report instrument used to assess for the presence of any pain-related TMD, with sensitivity and specificity ≥ 0.95 which is recommended for all patients in any clinical setting. A positive screen is followed by further evaluation to arrive at the specific TMD pain-related diagnoses.
DCTMD: AI Axis I Symptom questionnaire | 0 day
  Symptom questionnaire which assess pain characteristics as well as history of jaw noise, jaw locking, and headache.
DCTMD: AI Axis I Clinical Examination Form | 0 day
  Clinical Examination Form- The clinical examination includes provocation tests for TMJ arthralgia of pain with any jaw movement (ie, opening, lateral, and protrusive) and TMJ palpation. For myalgia, the tests include pain with opening jaw movements and palpation of the temporalis and masseter muscles.

SECONDARY OUTCOMES:
DCTMD: AI Axis II-Pain Drawing | 0 day
  Pain Drawing-pain drawing of the head, jaw, and body, and it allows the patient to report the location of all pain complaints
DCTMD: AI Axis II-Graded Chronic Pain (version 2) | 0 day
  Graded Chronic Pain (version 2) is a short, reliable, and valid instrument that assesses pain intensity and pain-related disability.10 The two GCPS subscales are: Characteristic Pain Intensity (CPI), which reliably measures pain intensity, with ≥ 50/100 considered "high intensity," and the pain-disability rating, which is based on number of days that pain interferes with activity and on extent of interference with social, work, or usual daily activities
DCTMD: AI Axis II-Jaw Functional Limitation Scale-8 (JFLS-8) | 0 day
  Jaw Functional Limitation Scale-8 (JFLS-8) which assesses global limitations across mastication, jaw mobility, and verbal and emotional expressionJFLS-8 is aimed to evaluate functional limitation of the jaw. The restriction due to TMD is indicated in eight items and these include changes in jaw mobility (item four), mastication (items 1-3), and verbal and emotional expression (items 5-8).Patient will asked to score between 0 and 10 according to the severity of the restriction. A higher score indicates more functional limitations.
DCTMD: AI Axis II-Patient Health Questionnaire (PHQ-4) | 0 day
  Patient Health Questionnaire (PHQ-4) is a short, reliable, and valid screening instrument for detecting "psychological distress" due to anxiety and/or depression in patients in any clinical setting.A cutoff of > 6, suggesting moderate psychological stress, should be interpreted as warranting observation, while a cutoff of > 9, suggesting severe psychological distress, should be interpreted as warranting either further assessment or referral
DCTMD: AI Axis II- Oral Behaviors Checklist (OBC) | 0 day
  Oral Behaviors Checklist (OBC), which assesses the frequency of oral parafunctional behaviors.

CONTACTS AND LOCATIONS:
Locations (1):
- Başak Çiğdem Karaçay, Yerköy, Yozgat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Goldstein RE, Auclair Clark W. The clinical management of awake bruxism. J Am Dent Assoc. 2017 Jun;148(6):387-391. doi: 10.1016/j.adaj.2017.03.005. PMID 28550845
- [Background] Poveda Roda R, Bagan JV, Diaz Fernandez JM, Hernandez Bazan S, Jimenez Soriano Y. Review of temporomandibular joint pathology. Part I: classification, epidemiology and risk factors. Med Oral Patol Oral Cir Bucal. 2007 Aug 1;12(4):E292-8. PMID 17664915
- [Background] Manfredini D, Lobbezoo F. Relationship between bruxism and temporomandibular disorders: a systematic review of literature from 1998 to 2008. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2010 Jun;109(6):e26-50. doi: 10.1016/j.tripleo.2010.02.013. PMID 20451831
- [Background] Lobbezoo F, Lavigne GJ. Do bruxism and temporomandibular disorders have a cause-and-effect relationship? J Orofac Pain. 1997 Winter;11(1):15-23. PMID 10332307
- [Background] Nakata A, Takahashi M, Ikeda T, Hojou M, Araki S. Perceived psychosocial job stress and sleep bruxism among male and female workers. Community Dent Oral Epidemiol. 2008 Jun;36(3):201-9. doi: 10.1111/j.1600-0528.2007.00388.x. PMID 18474052
- [Background] Guo H, Wang T, Niu X, Wang H, Yang W, Qiu J, Yang L. The risk factors related to bruxism in children: A systematic review and meta-analysis. Arch Oral Biol. 2018 Feb;86:18-34. doi: 10.1016/j.archoralbio.2017.11.004. Epub 2017 Nov 11. PMID 29149621
- [Derived] Cigdem Karacay B, Sahbaz T. Investigation of the relationship between probable sleep bruxism, awake bruxism and temporomandibular disorders using the Diagnostic Criteria for Temporomandibular Disorders (DC/TMD). Dent Med Probl. 2023 Oct-Dec;60(4):601-608. doi: 10.17219/dmp/158926. PMID 36651343